CLINICAL TRIAL: NCT05944224
Title: A Randomized, Open-label, Phase Ib/IIa Clinical Study to Evaluate the Efficacy and Safety of SPH4336 Monotherapy or in Combination With Cadonilimab in Patients With Advanced Solid Tumors, Including Advanced Well Differentiated/Dedifferentiated Liposarcoma.
Brief Title: A Study to Efficacy and Safety of SPH4336 Monotherapy or in Combination With Cadonilimab in Patients With Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPH4336-201
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SPH4336 (Experimental)
  Interventions: Drug: SPH4336
- Cadonilimab (Experimental)
  Interventions: Drug: Cadonilimab
- SPH4336+ Cadonilimab (Experimental)
  Interventions: Drug: SPH4336; Drug: Cadonilimab

INTERVENTIONS:
Drug: SPH4336 — SPH4336 Tablets ：Orally, 400mg once a day ; 28 days/cycle
  Arms: SPH4336; SPH4336+ Cadonilimab
Drug: Cadonilimab — Intravenous infusion, 6mg/Kg,28 days/cycle
  Arms: Cadonilimab; SPH4336+ Cadonilimab

SUMMARY:
This is a randomized, Open-label, Phase Ib/IIa study to evaluate the efficacy and safety of SPH4336 monotherapy or in combination with Cadonilimab in the patients with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in this study and sign informed consent.
2. Expected survival ≥3 months.
3. Patients with advanced solid tumors (including advanced Well differentiated/dedifferentiated liposarcoma) who cannot be treated by radical surgery/other local treatment.
4. According to RECIST v1.1, participants in the dose expansion phase must have at least one measurable lesion.
5. The laboratory test results meet the organ function requirements before starting the study treatment.
6. Prior to the start of the study treatment, the peripheral nerve toxicity of previous anti-tumor drug treatment had returned to ≤ grade 2, and other reversible toxic reactions had returned to ≤ grade 1, but hair loss/pigmentation and other effects were assessed by the investigator as beneficial to the subjects receiving the study treatment. The toxicity of the risk is not subject to this limitation.
7. Subjects agree to use effective contraception from the time they sign the informed consent to the last time they use the study drug.

Exclusion Criteria:

1. Taking anti-tumor traditional Chinese medicines at the time of signing the ICF.
2. Had undergone surgery prior to treatment and hasn't yet recovered from adverse effects of surgery.
3. Had a history of other malignancies before starting the study.
4. History of myocardial infarction, unstable angina pectoris, severe arrhythmia, and symptomatic congestive heart failure before the start of study treatment; NYHA Class ≥II; QTcF≥ 470 ms; LVEF≤ 50%.
5. Diseases affecting drug administration or gastrointestinal absorption before the start of the study and assessed by the investigators could not be included in the study.
6. Previous history of organ transplantation.
7. Before starting the study, HBsAg positive patients with HBV DNA > 500IU/ mL or 2500 copies /mL or the lower limit of the study center detection, or HCV antibody positive patients with HCV RNA positive, or known HIV-infected patients, or known active tuberculosis.
8. Accompanied by any other serious, progressive, or uncontrolled disease.
9. Subjects with a known history of immune-related adverse events that the investigator determined could not be included.
10. History of severe allergic disease, history of severe drug allergy, or known allergy to any component of the investigational product.
11. Women who are pregnant or breastfeeding.
12. Any other reason for which patients are ineligible for the study as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately 2 years
  From the start date of study treatment to the date of progression disease or death , whichever occurred first.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Approximately 2 years
  Tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1.
progression-free rate（PFR） | Approximately 2 years
  Proportion of subjects who were alive and free of disease progression from the first use of the investigational drug to 12 weeks.
Cmax | Approximately 2 years
  PK (Pharmacokinetics) parameters.
Tmax | Approximately 2 years
  PK (Pharmacokinetics) parameters.
Disease control rate (DCR) | Approximately 2 years
  DCR was defined as the percentage of patients who have achieved complete response, partial response and stable disease.
Duration of remission (DOR) | Approximately 2 years
  DOR was defined for participants who had an objective response as the time from the first occurrence of a documented unconfirmed response to the date of disease progression per RECIST v1.1 or death from any cause.
Overall Survival (OS) | Approximately 8 years
  Determination of the overall survival times of all patients.
Incidence of Adverse event | Approximately 2 years
  Safety and tolerability

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital，Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, He'nan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Central Hospital of Yongzhou, Yongzhou, Hunan
  - Liaoning Cancer Hospital & Institute, Shenzhen, Liaoning
  - Xijing Hospital, Xi’an, Shanxi
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang cancer Hospital, Hangzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin